CLINICAL TRIAL: NCT05269693
Title: A Brief Hope Intervention to Increase Hope Level and Decrease Stress Level of Parents With Children With Medical Complexity in the Community? A Pilot RCT
Brief Title: A BHI to Increase Hope Level and Stress Level of Parents With a CMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Winsome Lam, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPUSN
Record Dates: First submitted 2022-01-05; First posted 2022-03-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2022-02

CONDITIONS: Child With Cancer; Muscular Atrophy, Spinal; Child With Cerebral Palsy; Endocrine System Diseases
Keywords: Brief Hope Therapy; Parent; Children with medical complexity; stress
MeSH Terms: conditions — Muscular Atrophy, Spinal; Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: This is a single-blinded, pilot randomized controlled trial with two-armed repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Brief Hope Intervention group (Experimental): The BHI consisted of 4 one-on-one sessions: 2 (1 hr) face- to-face sessions, and 2 (30 min) telephone follow-up sessions in-between.
  Interventions: Other: Brief Hope Intervention
- wait-listed control group (No Intervention): Usual community care

INTERVENTIONS:
Other: Brief Hope Intervention — The BHI consisted of 4 one-on-one sessions: 2 (1 hr) face- to-face sessions, and 2 (30 min) telephone follow-up sessions
  Arms: the Brief Hope Intervention group

SUMMARY:
Being a parent of a child with medical complexity (CMC) poses an enormous stress because these CMC have a multisystem disease, a severe neurologic condition or cancer which may result in premature death. Parents may feel challenged, lacking in confidence and high level of stress when managing their daily caregiving activities and child's new symptom. Literature suggested that hope is believed to be the central agent in facilitating positive psychological change when parents are facing difficulties and feeling stress. Brief Hope Intervention (BHI) is an alternative method considered to be feasible in improving parental hope level meanwhile, decreasing their stress level associated with daily caregiving activities. The purpose of BHI is to help these parents to develop workable goals, and concentrate on problem solving skill along with achievable planned actions in order to terminate the stressors associated from the caregiving activities.

This proposed pilot randomized controlled trial will test the feasibility and preliminary effect of the BHI in term of increasing the level of hope meanwhile decreasing the stress level of parents with a CMC. Eligibility, recruitment rates, and attrition rates will be collected in percentage to evaluate the feasibility of the study. Content analysis will be adopted to analysis the qualitative feedback on the acceptability of BHI from the parents. A repeated-measures, two-group design will be used to evaluate the preliminary effects between intervention and wait-listed control groups by comparing Brief Hope Intervention and wait-listed control groups receiving usual community care for 64 randomly selected parents over a 1-month follow-up. The outcome measures include parental hope and stress level. They will be measured before intervention, immediately after intervention and one-month after intervention.

With positive outcomes found in this study, this intervention will be implemented in a larger scale to improve local psychological health service for parents with a CMC.

ELIGIBILITY:
Inclusion Criteria:

Parents of a CMC will be recruited via the special schools for the children with physical disabilities. The eligible criteria for parents are

1. one of the parent of a child with medical complexity aged 5-18,
2. able to communicate in Chinese and read Chinese,
3. willing to participate in face-to-face activities and a telephone follow-up,
4. alert and oriented, able to sustain approximately 1 hour of attention and interaction, and
5. able to be reached by phone.

Exclusion Criteria:

Parents are

1. a reported mental health disorder,
2. inability to communicate in Cantonese,
3. engaging in other Hope Therapy related to stress relief and hope enhancement, and
4. severe hearing deficit that prevented them from engaging in phone communication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | Week 4
  Enrollment and dropout rates will be calculated for each participant and summarized for all participants in the study
Intervention Delivery Rating Scale | Week 4
  5-point Likert scale for evaluating the useful level of intervention, ranging from 1 (not at all) to 5 (most).Higher scores mean more better outcome.
Change of Hope Level | Week 0, Week 4, Week 8
  State Hope Scale (Chinese version): consisting of 6 items. Each item is rated on a 8-point scale, with 1 = definitely false and 8 = definitely true. Higher scores mean higher hope level.
Change of Stress Level | Week 0, Week 4, Week 8
  Perceived Stress Scale (Chinese version): consisting of 14 items. Each item is rated on a 5-point scale, ranging from 1 (not at all) to 5 (extremely). Higher scores mean higher stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No